CLINICAL TRIAL: NCT06557772
Title: A Phase 2a/b, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of Subcutaneous Amlitelimab in Adult Patients With Nonresponsive Celiac Disease as an Adjunct to a Gluten-free Diet
Brief Title: A Phase 2a/b Study of the Efficacy and Safety of Subcutaneous Amlitelimab in Adults With Nonresponsive Celiac Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI17963; 2024-511213-38 (Registry Identifier: CTIS); U1111-1298-7193 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Coeliac Disease; Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Amlitelimab dose 1 + Gluten-free product (GFP) (Experimental): Amlitelimab SC as per protocol + GFP
  Interventions: Drug: Amlitelimab; Dietary Supplement: Gluten-free product (GFP)
- Amlitelimab dose 2 + GFP (Experimental): Amlitelimab SC as per protocol + GFP
  Interventions: Drug: Amlitelimab; Dietary Supplement: Gluten-free product (GFP)
- Amlitelimab dose 3 + GFP (Experimental): Amlitelimab SC as per protocol + GFP
  Interventions: Drug: Amlitelimab; Dietary Supplement: Gluten-free product (GFP)
- Amlitelimab dose 1 + SIGE (Experimental): Amlitelimab SC as per protocol + SIGE
  Interventions: Drug: Amlitelimab; Dietary Supplement: SIGE
- Placebo + GFP (Placebo Comparator): Placebo SC as per protocol + GFP
  Interventions: Drug: Placebo; Dietary Supplement: Gluten-free product (GFP)
- Placebo + SIGE (Placebo Comparator): Placebo SC as per protocol + SIGE
  Interventions: Drug: Placebo; Dietary Supplement: SIGE

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: SC injection
  Other Names: SAR445229
  Arms: Amlitelimab dose 1 + Gluten-free product (GFP); Amlitelimab dose 1 + SIGE; Amlitelimab dose 2 + GFP; Amlitelimab dose 3 + GFP
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: SC injection
  Arms: Placebo + GFP; Placebo + SIGE
Dietary Supplement: SIGE — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Amlitelimab dose 1 + SIGE; Placebo + SIGE
Dietary Supplement: Gluten-free product (GFP) — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Amlitelimab dose 1 + Gluten-free product (GFP); Amlitelimab dose 2 + GFP; Amlitelimab dose 3 + GFP; Placebo + GFP

SUMMARY:
This is a Phase 2a/b, randomized, double-blind, placebo-controlled, parallel-group, 6-arm study to evaluate the efficacy and safety of amlitelimab in adult participants with non-responsive celiac disease (NRCD) who are on a gluten free diet (GFD) with and without simulated inadvertent gluten exposure (SIGE).

The primary purpose of this study is to demonstrate the efficacy of subcutaneous (SC) amlitelimab in male and female participants (aged 18 to 75 years, inclusive) with NRCD. The study will assess the effect of amlitelimab when compared to placebo on gluten induced changes in the intestinal mucosa as measured by the villous height to crypt depth (Vh:Cd) ratio. The effect of amlitelimab on participant-reported celiac signs and symptoms along with the safety, tolerability, and pharmacokinetics of amlitelimab will also be studied.

Study details include:

The study duration will be up to 48 weeks (including a 16-week safety follow-up period) with 10 visits for participants who opt not to enter the optional long-term extension.

The study duration will be up to 172 weeks (including an 8-week safety follow-up period) with 22 visits for participants who enter the optional long-term extension.

The double-blind placebo-controlled treatment duration will be up to 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Participants with physician-diagnosed celiac disease with documented history of biopsy-proven celiac disease confirmed by medical records or physician statement.
* Participants who have self-reported attempt to maintain a GFD (and confirmed via questionnaire) for at least 12 consecutive months and must be willing to maintain their current diet for the duration of study participation.
* Participants have an adequate comprehension of a GFD as assessed by the Investigator.
* Participants willing to undergo all assessments in the protocol, including 2 esophagogastroduodenoscopies with duodenal biopsies.
* Participants who completed CDSD with ≥ 75% compliance from screening until randomization.
* During screening, participants must have at least one gastrointestinal symptom (i.e., diarrhea, abdominal pain, bloating, or nausea) of moderate or greater severity, as measured by the CDSD Gastrointestinal Domain, on at least 3 days out of any consecutive 7-day period considered by the investigator to be related to gluten exposure (i.e., due to celiac disease). The symptom can vary, but severity must be moderate or greater on three or more days. Participants must meet symptom criteria to undergo baseline esophagogastroduodenoscopy (EGD).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* A diagnosis of any severe complication of celiac disease, such as refractory celiac disease type 1 (RCD I) requiring immune suppressive medication, or type 2 (RCD II), enteropathy associated T-cell lymphoma (EATL), ulcerative jejunitis, or recent (within 12 months of screening) GI perforation.
* Presence of other active inflammatory GI disorders, including but not limited to the following: inflammatory bowel disease, eosinophilic esophagitis, diverticulitis, helicobacter infection, gastroenteritis or colitis, and microscopic colitis (requiring treatment) in the 6 months before screening. A history of treated erosive esophagitis is not an exclusion. Abnormalities found during baseline EGD or biopsy that are consistent with an inflammatory GI disorder other than celiac disease are exclusionary.
* Presence of other systemic autoimmune diseases including scleroderma, psoriatic or rheumatoid arthritis, and lupus. Participants with thyroid disease that has been well-controlled for at least 6 months, prior to screening, and participants with well-controlled type 1 diabetes (glycosylated hemoglobin < 9 % and no hospitalization or emergency room visit in the last 12 months for hyperglycemia or hypoglycemia) can be included per investigator judgement.
* Known or suspected severe enteric infection (viral, bacterial, or parasitic) within 6 months before screening. Severe enteric infection is defined as requiring a visit to the emergency room, hospitalization, or treatment with antibiotics or anti-infectives due to infection. Non-enteric viral infections, either resolved or well-controlled are not exclusionary.
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to screening (1 week in the event of superficial skin infections).
* Known history of or suspected significant current immunosuppression or hyposplenism, including history of invasive opportunistic or invasive helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Any malignancies or history of malignancies prior to enrollment (except for non-melanoma skin cancer that has been excised and completely cured for more than 5 years prior to enrollment).
* History of solid organ or stem cell transplant.
* Ongoing use, or use in the 3 months before screening, of medications known to cause villus abnormalities (eg, mycophenolate mofetil, azathioprine, methotrexate, olmesartan (other angiotensin receptor blockers are allowed), CTLA4 inhibitors, and PD-1/PD-L1 inhibitors).
* Ongoing chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) of more than 2 doses per week, except acetylsalicylic acid/aspirin ≤100 mg daily for prophylactic use.
* Any ongoing treatment with systemic immunosuppressants, systemic corticosteroids, or use of oral budesonide in the 12 weeks before screening.
* Ongoing use of over-the-counter digestive enzymes or supplements, other than lactase, including those for gluten digestion and oral pharmaceutical probiotic supplements. Probiotics in foods (e.g., yogurt) are permitted.
* Concurrent participation in any other clinical study, including non-interventional studies.
* Prior administration of investigational agents to treat celiac disease within 5 half-lives of any agent, or one year from any tolerogenic agent.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2029-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Villus Height to Crypt Depth Ratio (Vh:Cd) from baseline to Week 28 | Baseline to Week 28
  Change in Vh:Cd ratio.

SECONDARY OUTCOMES:
Change in Celiac Disease Symptom Diary (CDSD) Gastrointestinal (GI) symptom severity score | Baseline to Week 28
  The CDSD is a patient report outcome instrument that assesses common celiac symptoms (abdominal pain, bloating, tiredness, nausea, and diarrhea). GI symptom severity score ranges from 0-20 with higher score indicating more severe disease.
Percentage of participants who experienced treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) and adverse events of special interest (AESI) during the placebo-controlled treatment period and the long-term extension | Baseline to Week 168
Percentage of participants with potentially clinically significant abnormalities (PCSA) for vital signs and clinical laboratory assessments during the placebo-controlled treatment period and the long-term extension | Baseline to Week 168
Percentage of participants discontinued from study treatment due to TEAEs during the placebo-controlled treatment period and the long-term extension | Baseline to Week 168
Serum amlitelimab concentrations measured at prespecified timepoints | Baseline to Week 168
Incidence of antidrug antibodies (ADAs) of amlitelimab | Baseline to Week 168

CONTACTS AND LOCATIONS:
Locations (121):
- United States (37):
  - One of a Kind Clinical Research Center - Scottsdale- Site Number : 8400055, Scottsdale, Arizona
  - FOMAT Medical Research - inSite Digestive Health Care - Arcadia- Site Number : 8400052, Arcadia, California
  - Om Research - Lancaster - 15th Street West- Site Number : 8400001, Lancaster, California
  - United Medical Doctors - Los Alamitos- Site Number : 8400014, Los Alamitos, California
  - Om Research- Site Number : 8400010, Oxnard, California
  - Advanced Research Institute - Denver- Site Number : 8400048, Denver, Colorado
  - Medical Research Center of Connecticut- Site Number : 8400050, Hamden, Connecticut
  - Wellness Clinical Research - Miami Lakes - 8181 Northwest 154th Street- Site Number : 8400040, Miami Lakes, Florida
  - GI Pros- Site Number : 8400034, Naples, Florida
  - Center for Digestive Health- Site Number : 8400013, Orlando, Florida
  - GCP Clinical Research- Site Number : 8400007, Tampa, Florida
  - Treasure Valley Medical Research- Site Number : 8400006, Boise, Idaho
  - Hutchinson Clinic- Site Number : 8400020, Hutchinson, Kansas
  - University of Kansas Medical Center- Site Number : 8400041, Kansas City, Kansas
  - Boston Specialists- Site Number : 8400051, Boston, Massachusetts
  - Berkshire Medical Center- Site Number : 8400017, Pittsfield, Massachusetts
  - Gastroenterology Associates of Western Michigan - Wyoming- Site Number : 8400004, Wyoming, Michigan
  - Mayo Clinic in Rochester - Minnesota- Site Number : 8400049, Rochester, Minnesota
  - Washington University- Site Number : 8400025, St Louis, Missouri
  - Advanced Research Institute - Reno- Site Number : 8400036, Reno, Nevada
  - Sanmora Bespoke Clinical Research Solutions- Site Number : 8400015, East Orange, New Jersey
  - Allied Digestive Health - Middlesex Monmouth Gastroenterology- Site Number : 8400053, Freehold, New Jersey
  - M3 Wake Research- Site Number : 8400008, Raleigh, North Carolina
  - Thomas Jefferson University- Site Number : 8400056, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Providence- Site Number : 8400002, East Greenwich, Rhode Island
  - M3 Wake Research - Chattanooga- Site Number : 8400012, Chattanooga, Tennessee
  - Quality Medical Research- Site Number : 8400018, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Cedar Park- Site Number : 8400030, Cedar Park, Texas
  - MedCare Pharma - Houston - Cypress Creek Parkway- Site Number : 8400016, Houston, Texas
  - LinQ Research - Smith Ranch Road- Site Number : 8400028, Pearland, Texas
  - DM Clinical Research - Tomball- Site Number : 8400042, Tomball, Texas
  - Advanced Research Institute - Odgen- Site Number : 8400044, Ogden, Utah
  - Advanced Research Institute - Sandy - South 1300 East- Site Number : 8400046, Sandy City, Utah
  - Velocity Clinical Research - Salt Lake City- Site Number : 8400023, West Jordan, Utah
  - Gastroenterology Associates of Central Virginia- Site Number : 8400057, Lynchburg, Virginia
  - Clinical Research Partners - Richmond - Forest Avenue- Site Number : 8400011, Richmond, Virginia
  - GI Alliance - Tacoma- Site Number : 8400033, Tacoma, Washington
- Argentina (9):
  - Investigational Site Number : 0320007, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320010, Quilmes, Buenos Aires
  - Investigational Site Number : 0320008, San Isidro, Buenos Aires
  - Investigational Site Number : 0320012, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320009, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320002, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320003, Córdoba
- Australia (3):
  - Investigational Site Number : 0360002, Campbelltown, New South Wales
  - Investigational Site Number : 0360001, Mackay, Queensland
  - Investigational Site Number : 0360005, Box Hill, Victoria
- Belgium (2):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560001, Leuven
- Brazil (6):
  - Hospital Sao Rafael- Site Number : 0760005, Salvador, Estado de Bahia
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760006, Salvador, Estado de Bahia
  - Chronos Pesquisa Clínica- Site Number : 0760002, Brasília, Federal District
  - Hospital Moinhos de Vento- Site Number : 0760004, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Praxis Pesquisas Medicas- Site Number : 0760008, Santo André, São Paulo
- Canada (2):
  - Investigational Site Number : 1240001, Vancouver, British Columbia
  - Investigational Site Number : 1240002, Victoria, British Columbia
- Chile (6):
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Concepción, Región del Biobío
  - Investigational Site Number : 1520005, Talcahuano, Región del Biobío
- Czechia (5):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030006, Havířov
  - Investigational Site Number : 2030005, Klatovy
  - Investigational Site Number : 2030001, Prague
  - Investigational Site Number : 2030003, Prague
- Finland (3):
  - Investigational Site Number : 2460002, Helsinki
  - Investigational Site Number : 2460003, Tampere
  - Investigational Site Number : 2460001, Turku
- France (2):
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500001, Paris
- Germany (4):
  - Investigational Site Number : 2760006, Berlin
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760001, Halle
  - Investigational Site Number : 2760002, Mainz
- Greece (2):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Athens
- Israel (6):
  - Investigational Site Number : 3760002, Afula
  - Investigational Site Number : 3760006, Beersheba
  - Investigational Site Number : 3760004, Jerusalem
  - Investigational Site Number : 3760003, Petah Tikva
  - Investigational Site Number : 3760007, Ramat HaSharon
  - Investigational Site Number : 3760001, Rehovot
- Italy (3):
  - Ospedale Maggiore Policlinico Milano-Site Number : 3800002, Milan, Milano
  - Azienda Ospedaliera di Padova-Site Number : 3800004, Padua, Padova
  - Ospedale di Cisanello-Site Number : 3800003, Pisa
- Netherlands (2):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280002, Arnhem
- Poland (4):
  - Investigational Site Number : 6160004, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160005, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160002, Warsaw, Masovian Voivodeship
- Slovakia (3):
  - Investigational Site Number : 7030001, Košice
  - Investigational Site Number : 7030003, Nitra
  - Investigational Site Number : 7030004, Šahy
- Spain (9):
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240009, Chiclana de la Frontera, Cádiz
  - Investigational Site Number : 7240011, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240002, Seville, Sevilla
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240004, Málaga
  - Investigational Site Number : 7240008, Seville
  - Investigational Site Number : 7240010, Seville
- Sweden (4):
  - Investigational Site Number : 7522001, Linköping
  - Investigational Site Number : 7521001, Mölndal
  - Investigational Site Number : 7520003, Stockholm
  - Investigational Site Number : 7520001, Uppsala
- Turkey (Türkiye) (7):
  - Investigational Site Number : 7920004, Antalya
  - Investigational Site Number : 7920003, Gaziantep
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920007, Izmir
  - Investigational Site Number : 7920001, Mersin
  - Investigational Site Number : 7920005, Sanliurfa
  - Investigational Site Number : 7920002, Zonguldak
- United Kingdom (2):
  - Investigational Site Number : 8260001, Oxford, Oxfordshire
  - Investigational Site Number : 8260002, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI17963 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26057&tenant=MT_SNY_9011